CLINICAL TRIAL: NCT03481426
Title: Workplace Interventions Supporting Employees to Continue at Work: Participatory Actions Organized by OH Physiotherapist
Brief Title: The Effect of Workplace Interventions on the Treatment of Low-back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Institute of Occupational Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ESormunen
Record Dates: First submitted 2017-11-06; First posted 2018-03-29 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Back Pain
Keywords: musculoskelelal disorder; occupational health service
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Workplace intervention group (Experimental): Workers with back problems receive both information/advice and participatory workplace intervention organized by Occupational Health Physioterapist.
  Interventions: Other: Workplace intervention
- Information and advice group (No Intervention): Workers with back problems receive only information / advice by Occupational Health Physiotherapist, not the workplace intervention.

INTERVENTIONS:
Other: Workplace intervention — The study contains normal services of occupational health. Both intervention groups are based on voluntary will, and the normal care and services are guaranteed. In the intervention group new working method which improve co-operation between occupational health services and workplaces.
  Arms: Workplace intervention group

SUMMARY:
The study evaluates the effect of workplace interventions on work ability promotion among workers with back problems. The half of participant will receive Information, advice and guidance for back problems in addition to participatory workplace actions organized by Occupational Health Physiotherapist. The other half will receive only Information, advice and guidance without workplace intervention.

DETAILED DESCRIPTION:
Musculoskeletal symptoms, especially back pain, account for the majority of days lost.

In order to enhance the health and working careers of people with MSD, it is important that work can be arranged in such a way that they can remain in work life despite MSD.In the field of work ability promotion, various stakeholders; the worker, employer, professionals in occupational health services (OHS) interact to optimize actions and practices to prevent absences from work and promote remaining at work. This study aims to investigate participatory working practices and modles of co-operation among OHS and workplaces.

ELIGIBILITY:
Inclusion Criteria:

* Back pain for at least two weeks or frequently occuring periods within the past 12 months

Exclusion Criteria:

* Back problems with forcoming surcical operation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
work ability | through study completion, up to 12 months
  The present self estimated work ability versus the life time best (0-10)

SECONDARY OUTCOMES:
intensity of pack pain | through study completion, up to 12 months
  The present self estimated back pain, no pain - the worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Erja Sormunen, PhD, Principal Investigator — Finnish Institute of Occupational Health
Locations (1):
- Finnish Institute of Occupational Health, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
All the collected data and study results are analyzed anonymous and are kept under the control of the Project group. All the personal data and information of the participants are kept under the control of the Project researchers.